CLINICAL TRIAL: NCT04941924
Title: A Pilot Multicentre Prospective Randomised Controlled Trial Comparing the Safety and Efficacy of Intraductal Radio-frequency Ablation (ID-RFA) Using Starmed's Temperature Controlled ELRA™ Probe Plus Biliary Stenting Versus Biliary Stenting Alone for the Treatment of Malignant Biliary Obstruction.
Brief Title: The ID- RFA Trial: A Trial of Intraductal Radio-frequency Ablation (ID-RFA) Plus Biliary Stenting Versus Biliary Stenting Alone for the Treatment of Malignant Biliary Obstruction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals Dorset NHS Foundation Trust (Other Government)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 274029
Record Dates: First submitted 2021-06-10; First posted 2021-06-28 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-05

CONDITIONS: Malignant Biliary Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Biliary stenting plus radio-frequency ablation of the bile duct
  Interventions: Procedure: Intraductal Radio-Frequency Ablation; Device: Biliary Stent Placement
- Control (Active Comparator): Biliary stenting alone
  Interventions: Device: Biliary Stent Placement

INTERVENTIONS:
Procedure: Intraductal Radio-Frequency Ablation — The electrode employed in this study is the STARmed ELRA™ (Endo Luminal Radiofrequency Ablation) electrode; this is a CE marked device. The selected electrode will be connected to the VIVA™ Combo generator (also a CE marked device) and advanced over the guide wire.
  The power of the generator should be set at either 7 or 10 W depending on the electrode used per manufacturer instructions. An ablation should then be applied at a temperature of 70 to 80℃ for 2 minutes. For longer length strictures or stent occlusions, the RFA probe is withdrawn from proximal to distal in a step by step fashion in respect to the access method used.
  Arms: Intervention
Device: Biliary Stent Placement — Taewoong Niti-S™ LCD Biliary stents (CE marked uncovered self-expanding metal stents) placed according to standard local practice.

SUMMARY:
Cancers of the liver, pancreas and gall bladder can partially or fully block the bile duct leading to jaundice. Where these tumours are inoperable, maintaining adequate bile duct drainage is an important factor in survival, both as jaundice itself can ultimately be fatal and because and because it can prevent the administration of chemotherapy. The current standard care is the placement of a stent and possible manual 'trawling' in an attempt to clear the blockage. But these stents often become blocked by tumour ingrowth requiring reintervention. However it may not be safe to do so at this point.

Intraductal radiofrequency ablation (IDRFA) uses heat energy both to 'necrose' the tumour tissue in attempt to slow ingrowth in the channels before inserting stents and to clear blocked stents. There is some evidence that this increases the length of time for the stents to become blocked or with secondary benefits to quality of life and survival however long term data from within the NHS setting is lacking. A full trial is not currently feasible therefore a pilot study is to be conducted to help inform the design of a full trial.

This study will randomise patients attending with malignant biliary obstruction in a 1:1 ratio to receive either intraductal radiofrequency a. Participants will be recruited through the standard clinical pathway (i.e it will be offered to all potentially eligible patients) over a period of 12 months. Participants will be monitored for a period of up to 12 months for survival, stent blockage, symptoms, resource use, quality of life and adverse reactions.

The study will be conducted between Royal Bournemouth Hospital and The Christie, both cancer care centres experienced in the management of these conditions, stent placement and radiofrequency ablation.

DETAILED DESCRIPTION:
This trial will follow a multicentre randomised controlled trial design.

Patients will be recruited by the standard clinical pathway. Patients with these cancers will be under the care of the oncology team, this may be a new referral (fast-track cancer) or ongoing care. If they are symptomatic of potential biliary obstruction (jaundiced) they will undergo an ultrasound and/or CT scan to determine the cause. In the case of fast-track referrals a biopsy will be taken where possible to confirm diagnosis. If these investigations confirm biliary obstruction the case will be referred to the upper gastrointestinal cancer multidisciplinary team for review. In the case of newly diagnosed patients, if the tumour is resectable and the patient is fit for surgery then the patient will be referred to the appropriate surgical team. In newly diagnosed patients the patient may also be referred to the medical oncology team for consideration for chemotherapy or other systemic treatment however this will generally occur after the procedure being studied as such cases are generally 'emergencies' with reliving the obstruction being the most important prognostic factor in the short term.

Patients unsuitable or unwilling for surgery will then be reviewed by the interventional radiology/endoscopy team, either in clinic as an outpatient or on the ward as an inpatient depending on the nature of their case. If as an inpatient this is often performed in conjunction with the oncology team. Treatment options will be discussed with the patient including biliary stenting and at this point the trial will be introduced. The patient will be provided with written information and given the opportunity to ask any questions they may have about the trial. If the original CT imaging does not provide a clear indication of the location of the obstruction the patient will also be referred for magnetic resonance cholangiopancreatography.

Once given sufficient time to consider the study the patient will be reviewed again to make a decision on the course of treatment they would like to take and at this point if willing written informed consent will be taken. The duration of this period will be determined by the nature of the case however adequate time will be given. The results from the previous work-up and any other relevant medical history will be reviewed alongside a clinical assessment a by the investigator to confirm eligibility. This will be entered onto the eCRF prior to randomisation.

Once the patient has been confirmed as eligible and entered into the trial the procedure will be arranged. If the participant is suitable for stenting but not eligible for the trial this will be performed outside the trial. Prior to the procedure blood samples will be collected for Full Blood Count ,liver profile, renal profile and clotting analyses. The participant will also complete two baseline quality of life questionnaires and baseline symptom scores will be recorded.

The patient will then undergo intraductal radiofrequency ablation and biliary stenting. In accordance with local practice, at Bournemouth the approach used will be determined by the nature of the case, where the obstruction is below the cystic duct and the patient is suitable for general anaesthetic endoscopic retrograde cholangiopancreatography will be used. Where the obstruction is above the cystic duct or at the hilium, the participant has altered gastrointestinal anatomy or the participant is unsuitable for general anaesthetic, percutaneous transhepatic cholangiography will be used. At the Christie all procedures will use the latter approach. The procedure used will be the same for primary biliary obstruction and biliary stent occlusion. The participant will be discharged once deemed medically fit.

The participant will be asked to attend 2 follow-up visits, at one week and 1 month following the procedure. At this visit they will undergo a clinical review of their symptoms and any complications from the procedure. A blood sample will be collected and they will be asked to complete the quality of life questionnaires again. Participants will also be asked these quality of life questionnaires at home at 2,3, 6 and 12 months post procedure alongside an additional short questionnaire evaluating their symptoms and healthcare use. After the 1 month visit they be followed up as per standard care by the oncology team and any relevant information will be collected for the study. The participant will be monitored for stent occlusion and any relevant clinical findings recorded if this is suspected. This will be confirmed by at least 1 investigation in accordance with standard practice. The participant may be referred for further stenting which will be recorded in the patients eCRF. At this point trial follow up (questionnaires and recording of routine care visits) will terminate however the patient will continue to monitored for survival. Otherwise patients will undergo a CT scan at 12 months post procedure to evaluate stent patency and monitored until death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-85 years;
2. A cytological/histological or radiological diagnosis of inoperable HPB malignancy;
3. MDT review confirming inoperability.

   -Patients who have declined surgery will also be considered for the study.
4. Medically fit to undergo procedure in opinion of the investigator.

Exclusion Criteria:

1. Unable to provide free informed consent within 7 days;
2. ECOG performance status 3 or 4;
3. Life expectancy <1 months;
4. Prior investigational drugs within last 30 days;

   - Patients who have already commenced approved chemotherapy regimens are not excluded from the study.
5. Patients with clinically significant ascites;
6. Patients with CNS metastases;
7. Major surgery within last 30 days;
8. Patients with active sepsis or encephalopathy;

   - Patients may present with biliary sepsis prior to diagnosis. Inclusion of such a patient can be considered once biliary sepsis has been managed as per local Trust guidance.
9. Evidence of spontaneous bacterial peritonitis or renal failure;
10. Pregnant or lactating women;

    - Females of childbearing potential will undergo a blood pregnancy test to confirm they are not pregnant within 7 days prior to randomisation.
11. Unstable angina, heart disease or diabetes;
12. Intractable severe blood coagulation dysfunction;
13. Fitted with implantable pacemaker, implantable cardioverter/defibrillator or other active implant;
14. Unable to understand the study information or unable to complete the outcome questionnaires (in English);
15. Un-willing or un-able to comply with all protocol requirements including scheduled visits, treatment plans, laboratory tests and other study procedures;
16. Medically un-fit to undergo procedure in opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 12 months
  The average number of participants consented per month.

SECONDARY OUTCOMES:
Retention rate | 12 months
  The percentage of overall patients who consent to the trial and are not withdrawn either by their own choice or clinicians. Death does not constitute withdrawal.
Assessment Adherence | 12 months
  The percentage of protocol defined assessments completed in accordance with the protocol for patients who are alive and remain within the study at that point.
Intervention free survival | 12 months
  The time in days between receiving the intervention and either repeated stenting due to occlusion or death.
Overall survival | 12 months
  The number of days from receiving the intervention to patient death.
Stent Patency | 12 months
  The number of days from the procedure to Stent Occlusion confirmed by imaging or biochemistry (blood tests).
Increase in ductal caliber following intervention | Day 0
  Determined by comparison of imaging collected during the index procedure pre intervention and following both RFA for the experimental arm, and following stent placement for both arms. This will be measured at the narrowest stricture point.
Restoration of Biliary flow following intervention as determined by imaging during procedure | Day 0
Rates of cholangitis related to stent dysfunction | 12 months
  The percentage of patients who experience such an event.
EQ-5D-5L quality of life questionnaire | Pre procedure, and at 1 week and 1, 2, 3, 6 and 12 months post procedure.
  Participants will be asked to complete the EQ-5D-5L quality of life questionnaire, and index value calculated according to the user guide.
QLQ-C30 quality of life questionnaire | Pre procedure, and at 1 week and 1, 2, 3, 6 and 12 months post procedure.
  Participants will be asked to complete the QLQ-C30 quality of life questionnaire including an module determined by cancer type; QLQ-BIL21 (Cholangiocarcinoma and Gallbladder Cancer), QLQ-HCC18- (Hepatocellular Carcinoma) or QLQ-PAN26 (Pancreatic Cancer).
Symptom Score | Pre procedure, and at 1 week and 1, 2, 3, 6 and 12 months post procedure.
  Participants will be assessed for jaundice, nausea, bloating and abdominal pain, if present this will be graded according to CTCAE v5.0 criteria.
Serum bilirubin (in μmol/L) | At baseline, within 24 hours before the procedure, within 24 hours after, and at 1 week and 1, 2, 3, 6 and 12 months post procedure.
Alkaline phosphatase (in iu/L) | At baseline, within 24 hours before the procedure, within 24 hours after, and at 1 week and 1, 2, 3, 6 and 12 months post procedure.
Alanine transaminase (in iu/L) | At baseline, within 24 hours before the procedure, within 24 hours after, and at 1 week and 1, 2, 3, 6 and 12 months post procedure.
International normalized ratio | At baseline, within 24 hours before the procedure, within 24 hours after, and at 1 week and 1, 2, 3, 6 and 12 months post procedure.
  Calculated from prothrombin time,

OTHER OUTCOMES:
Resource Use - Operative Room Time | During Procedure
  This will be recorded from when the patient first enters the radiology or endoscopy room to the time that they leave. This will be used to make an assessment of facility and staff costs.
Resource Use - Admission Length | During admission, expected within range Day -7 to Day +14
  The total time that the patient is admitted for the procedure including recovery and prolonged admission due to complications. This will be used to make an assessment of facility and staff costs.
Resource Use - Hospital Recovery Time | During admission, Day 0 up to Day +14 (expected)
  The total time that the patient is admitted from procedure completion to full discharge. This will be used to make an assessment of facility and staff costs.
Resource Use - Quantity and details of single use devices and non-medicinal supplies utilised during procedure | During procedure
  Any single use items used in the procedure will be recorded including; RFA catheter, balloon catheter, stents and any other ancillary supplies. This will be used calculate the cost of the equipment used in the procedure.
Resource Use - Medication Usage (name, dosage, frequency and duration of) | During admission
  All medications used during the patient admission including prophylactic medication and that used to manage any adverse events. This may include parenteral fluids and blood products. Any medication that the participant routinely received prior to entry to the trial will be not be included. This will be used calculate the cost of the medication administered during admission.
Resource Use - Subsequent healthcare attendances (type, number and duration of) | through study completion, up to 12 months
  Any clinic visits, admissions and subsequent procedures relating to the trial indication or complications of the intervention that the patient undergoes in the 12 month trial period. This will be used to make an assessment of facility and staff costs.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.uhd.nhs.uk/hospitals-poole/services/96-services/joint-service/research